CLINICAL TRIAL: NCT05312047
Title: Urinary Continence Status After Vaginal Surgery for Prolapse Correction.
Brief Title: Continence After Vaginal Prolapse Surgery
Status: Completed | Type: Observational
Sponsor: Hospital Universitari Vall d'Hebron Research Institute (Other)
Collaborators: Consorci Sanitari de Terrassa (Other); Parc Taulí Hospital Universitari (Other); Hospital de Viladecans (Other); Hospital Universitari de Bellvitge (Other); Hospital d'Igualada (Other); Hospital de Mataró (Other); Fundació Hospital de l'Esperit Sant (Unknown); Germans Trias i Pujol Hospital (Other); Hospital Santa Caterina (Unknown); Hospital de Granollers (Other); Hospital del Mar (Other); Hospital Universitari Joan XXIII de Tarragona. (Other); Fundació Institut de Recerca de l'Hospital de la Santa Creu i Sant Pau (Other)
Responsible Party: Sponsor
Other Study IDs: PR(AMI)631-2021
Record Dates: First submitted 2022-03-17; First posted 2022-04-05 (Actual); Last update posted 2025-12-31 (Actual); Status verified 2025-12

CONDITIONS: Pelvic Organ Prolapse; Urinary Incontinence
Keywords: Pelvic organ prolapse; Surgery; Urinary incontinence; Stress urinary incontinence; Urge-urinary incontinence
MeSH Terms: conditions — Pelvic Organ Prolapse; Urinary Incontinence; Urinary Incontinence, Stress; Urinary Incontinence, Urge

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Pelvic organ prolapse surgery — Vaginal surgery of any compartment for pelvic organ prolapse

SUMMARY:
Urinary incontinence after surgical correction of pelvic organ prolapse (POP) could occur. This is a condition that decreases both patients' satisfaction and quality of life. Reports on the prevalence of urinary incontinence after POP surgery are controversial. Concomitant surgery for incontinence could reduce this prevalence, whereas it increases treatment costs and the likelihood of surgical complications. Therefore, it is of paramount importance to know the exact prevalence of urinary incontinence after POP surgery in our population and the potential risk factors associated with this condition.

ELIGIBILITY:
Inclusion Criteria:

* Women who will undergo vaginal surgery for pelvic organ prolapse.

Exclusion Criteria:

* Inability to give consent to the study.

Ages: 18 Years to 99 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients referred to different Spanish-Catalan hospitals with symptomatic pelvic organ prolapse who are candidates for surgical correction of their POP.
Sampling Method: Non-Probability Sample
Enrollment: 609 (Actual)
Dates: Start 2022-04-04 (Actual); Primary Completion 2025-09-19 (Actual); Study Completion 2025-09-19 (Actual)

PRIMARY OUTCOMES:
Stress urinary incontinence (SUI). | 1 year after surgery.
  A "Yes" response to any of three questions on the spanish version of the Pelvic Floor Distress Inventory (PFDI) stress incontinence subscale regarding leakage with coughing, sneezing, or laughing; physical exercise; and lifting or bending over (PFDI questions 20, 21 and 22) .
Urgency urinary incontinence (UUI). | 1 year after surgery.
  A "Yes" response to PFDI question 19, "usually experiences urine leakage associated with a feeling of urgency, that is, a strong sensation of needing to go to the bathroom".

SECONDARY OUTCOMES:
Incontinence severity | 1 year after surgery.
  Both SUI and UII severity will be assessed using the spanish versions of the Sandvik's severity index and the International Consultation on Incontinence Questionnaire Short Form (ICIQ-SF).
Patients' satisfaction with the procedure. | 1 year after surgery.
  Assessed with the Patient Impression of Improvement (PGI-I) form.

CONTACTS AND LOCATIONS:
Overall Officials: Marina Catalan, MD, Principal Investigator — Vall d'Hebron Barcelona Hospital Campus; Jordi Sabadell, MD, Study Director — Vall d'Hebron Barcelona Hospital Campus
Locations (14):
- Spain (14):
  - Hospital Germans Trias i Pujol, Badalona, Barcelona
  - Vall d'Hebron Barcelona Hospital Campus, Barcelona, Barcelona
  - Hospital General de Granollers, Granollers, Barcelona
  - Hospital d'Igualada, Igualada, Barcelona
  - Hospital General de l'Hospitalet, L'Hospitalet de Llobregat, Barcelona
  - Hospital Universitari de Bellvitge, L'Hospitalet de Llobregat, Barcelona
  - Parc Taulí Hospital Universitari, Sabadell, Barcelona
  - Hospital de l'Esperit Sant, Santa Coloma de Gramenet, Barcelona
  - Consorci Sanitari de Terrassa, Terrassa, Barcelona
  - Hospital de Viladecans, Viladecans, Barcelona
  - Hospital de Sant Pau, Barcelona
  - Hospital del Mar, Barcelona
  - Hospital Santa Caterina, Girona
  - Hospital Joan XXIII, Tarragona

IPD SHARING:
Plan to Share IPD: Undecided